CLINICAL TRIAL: NCT07115394
Title: EEG Measurements to Capture DBS-induced Electric Potentials
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: University of Twente (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-101217-BO-ff_1; 101116047 (Other Grant/Funding Number: European Research Council)
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Deep Brain Stimulation; Parkinson's Disease
Keywords: deep brain stimulation; EEG; electric potential

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EEG measurement during DBS: Different DBS conditions can include the individual bilateral therapeutical DBS settings, unilateral versions of these setting, unilateral single segment use of these settings or unilateral low frequency (15-30 Hz) DBS. EEG measurements with a 4-channel analog EEG amplifier (Digitimer EEG).
  Interventions: Other: EEG recording

INTERVENTIONS:
Other: EEG recording — EEG will be recorded at high sampling rate

SUMMARY:
To measure the electric fields induced by DBS (deep brain stimulation) on the scalp and to improve electric field simulations, the investigators will measure EEG (electroencephalography) measurements with high sampling rates (>100 kHz). The investigators hypothesize that we can improve electric field simulations of DBS by validating and calibrating the simulations based on EEG measurements at high sampling rates (>100 kHz).

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent by the patient
* Age 35 - 85
* patient groups: Parkinson's disease, essential tremor, dystonia
* >3 months after surgery for DBS

Exclusion Criteria:

none.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients implanted with deep brain stimulation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Electric potential at the EEG locations | during DBS
  The investigators will extract the DBS pulses from the EEG data and check the distribution of the electric potentials as seen in simulations based on individual MRI and CT images. Parameters of the simulation pipeline (e.g. conductances) will be adjusted so that the simulation models fit the data.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided